CLINICAL TRIAL: NCT00052676
Title: French Randomized Sentinel Node Multicentric Study
Brief Title: Technetium Tc 99m Sulfur Colloid and Blue Dye In Detecting Sentinel Lymph Nodes in Patients With Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Paul Strauss (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Diagnostic
Other Study IDs: STRAUSS-FRANSENOD; CDR0000258612 (Registry Identifier: PDQ (Physician Data Query)); EU-20214
Record Dates: First submitted 2003-01-24; First posted 2003-01-27 (Estimated); Last update posted 2013-05-15 (Estimated); Status verified 2007-09

CONDITIONS: Breast Cancer
Keywords: stage I breast cancer; stage II breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — iso-sulfan blue; Sentinel Lymph Node Biopsy; Technetium Tc 99m Sulfur Colloid

INTERVENTIONS:
Drug: patent blue V dye
Procedure: radionuclide imaging
Procedure: sentinel lymph node biopsy
Radiation: technetium Tc 99m sulfur colloid

SUMMARY:
RATIONALE: It is not yet known whether injecting technetium Tc 99m sulfur colloid and blue dye near the tumor is more effective than injecting them near the nipple in identifying sentinel lymph nodes in patients with stage I or stage II breast cancer.

PURPOSE: Randomized diagnostic trial to compare the effectiveness of injecting technetium Tc 99m sulfur colloid and blue dye near the tumor with that of injections around the nipple in detecting sentinel lymph nodes in patients who have stage I or stage II breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the optimal mode of injection (peritumoral vs periareolar) of patent blue V dye and technetium Tc 99m sulfur colloid in patients with stage I or II breast cancer undergoing sentinel lymph node identification.
* Determine the reduction of morbidity associated with breast cancer surgery, in terms of local control and survival, in patients undergoing sentinel lymph node identification with these drugs.
* Determine the evolution of disease in patients who have undergone this procedure and do not show histological invasion of the sentinel lymph node.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to participating center. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive peritumoral injections of patent blue V dye and technetium Tc 99m sulfur colloid.
* Arm II: Patients receive periareolar injections as in arm I. Patients in both arms showing histological metastasis of the sentinel lymph node or without identification of the sentinel lymph node undergo standard axillary lymph node dissection.

Patients are followed for disease evolution.

PROJECTED ACCRUAL: A total of 450 patients (225 per arm) will be accrued for this study within 2-2.5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed invasive breast cancer

  * T0, T1, or T2 no greater than 3 cm, N0
  * Amenable to surgery
* No inflammatory breast cancer
* No ductal cancer in situ or multicentric invasive ductal cancer
* No nipple/areola or central breast cancer (at least 2 cm from areola)
* No metastatic disease
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age

* Over 18

Sex

* Not specified

Menopausal status

* Not specified

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

Other

* Not pregnant
* Negative pregnancy test
* No known allergy or intolerance to patent blue V dye

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* No prior surgery for cancer

Other

* No prior neoadjuvant treatment for cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-10; Study Completion 2007-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Francois Rodier, MD, Study Chair — Centre Paul Strauss
Locations (7):
- France (7):
  - Clinique Tivoli, Bordeaux
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre Leon Berard, Lyon
  - Institut J. Paoli and I. Calmettes, Marseille
  - Centre Regional Rene Gauducheau, Nantes-Saint Herblain
  - Centre Paul Strauss, Strasbourg
  - Institut Claudius Regaud, Strasbourg

REFERENCES:
- [Result] Rodier JF, Velten M, Wilt M, Martel P, Ferron G, Vaini-Elies V, Mignotte H, Bremond A, Classe JM, Dravet F, Routiot T, de Lara CT, Avril A, Lorimier G, Fondrinier E, Houvenaeghel G, Avigdor S. Prospective multicentric randomized study comparing periareolar and peritumoral injection of radiotracer and blue dye for the detection of sentinel lymph node in breast sparing procedures: FRANSENODE trial. J Clin Oncol. 2007 Aug 20;25(24):3664-9. doi: 10.1200/JCO.2006.08.4228. Epub 2007 May 7. PMID 17485709